CLINICAL TRIAL: NCT00237042
Title: Hormonal Cycles in Women: Effects on TMD Pain & Symptoms
Brief Title: Managing Temporomandibular Disorder (TMD) Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Dr. Linda LeResche, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27729-D; R01DE016212 (NIH); 5R01DE016212 (NIH); NIDCR-16212 (Other Grant/Funding Number: National Institute of Dental and Craniofacial Research (NIDCR))
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-06

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Disorders; TMJ Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Self-Management; Ethinyl Estradiol; Levonorgestrel; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Self Management (Active Comparator): Dental hygienist-delivered pain self-management treatment
  Interventions: Behavioral: Self Management
- Targeted Self Management (Experimental): Dental hygienist-delivered pain self-management treatment with a focus on menstrual cycle-related changes in pain and other symptoms
  Interventions: Behavioral: Targeted Self Management
- Continuous Oral Contraceptives (Experimental): Oral contraceptive (20 mcg ethinyl estradiol and 100 mcg levonorgestrel) taken daily for 6 months with no "spacer pills."
  Interventions: Drug: 20 mcg ethinyl estradiol and 100 mcg levonorgestrel

INTERVENTIONS:
Behavioral: Self Management — Two 1.5-hour in-person sessions and 6 10-15-minute telephone calls delivered by a dental hygienist, trained and supervised by a clinical psychologist. Structured, manual-based treatment based on standard cognitive-behavioral pain therapies and self-management interventions for chronic TMD pain. Sessions included education about the biopsychosocial model of chronic pain, TMD etiology and treatments, and the rationale for self-management; relaxation and stress management training; discussion of the role of stress and emotions as potential factors exacerbating and maintaining TMD symptoms; instruction and practice in self-monitoring of symptoms to identify factors that might be helpful to modify through self-care methods; practice of dentist-prescribed self-care treatments; and discussion of strategies to maintain gains and prevent relapse.
  Arms: Self Management
Behavioral: Targeted Self Management — Self management as described above. However, the intervention also included education about the potential effects of hormones on TMD pain, instructions to monitor the association of pain and other symptoms with menstrual cycle changes, and planning for times in participants' menstrual cycles when symptoms might increase. Participant contacts were timed according to each participant's menstrual cycle.
  Arms: Targeted Self Management
Drug: 20 mcg ethinyl estradiol and 100 mcg levonorgestrel — Combination pill (20 mcg ethinyl estradiol and 100 mcg levonorgestrel) taken daily for 6 months.
  Other Names: Aviane
  Arms: Continuous Oral Contraceptives

SUMMARY:
The purpose of this study is to determine whether treatments targeted to the hormonal factors and the cyclicity of TMD symptoms associated with the menstrual cycle are more effective in relieving TMD pain and symptoms than standard self management treatment.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are a group of painful conditions involving the muscles of mastication and the temporomandibular joint. These pain problems are about twice as common in women as in men in the community, and prevalence peaks during the reproductive years. The etiology of TMD pain is unknown, but psychological stress, depression and the presence of other somatic complaints have been shown to influence the course of these disorders. Prior research suggests that female reproductive hormones may also influence TMD pain. Specifically, normally cycling women with TMD experience rising levels of TMD pain pre-menstrually during a time of precipitous drop in estrogen and show peak TMD pain during menses. Interestingly, a secondary peak of TMD pain occurs at about the time of ovulation, another phase corresponding to rapid estrogen change. These data demonstrate a systematic relationship between levels of TMD pain and phases of the menstrual cycle. The proposed clinical trial will manipulate the behavioral and hormonal factors that are hypothesized to influence TMD pain, comparing the effects of:

* a continuous oral contraceptive intervention designed to suppress menses and stabilize the hormonal environment;
* a self-management intervention focused on and timed to the chronobiology of TMD symptoms across the menstrual cycle; and
* a usual self-management intervention not timed to biological events. The aims of this clinical trial are to shed light on the mechanisms underlying the cyclic nature of TMD pain and symptoms in women, as well as to determine which treatment modality results in the greatest improvement in TMD pain and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* TMD Pain Diagnosis as determined by enrollment exam at the University of Washington
* Menstruate on a regular basis
* Not planning to become pregnant during the next 6 months

Exclusion Criteria:

* Drug or alcohol abuse
* Current smoker and 35 years of age at any time during the study
* Live further than 1 hour driving distance from the University of Washington, Seattle campus
* Psychiatric disability

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2005-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda LeResche, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited 10/05-06/09. Study participants were recruited from patients seeking care at the University of Washington Orofacial Pain Clinic and by advertising.
Pre-assignment Details: Run-in period: Study participants completed daily diaries of pain and other symptoms for one menstrual cycle prior to randomization. Only participants who returned completed diaries for at least 85% of the requested days were eligible for randomization. 191/252 enrolled subjects were randomized.
Groups:
- Targeted Self Management: Self management as described for the first arm. However, the intervention also included education about the potential effects of hormones on TMD pain, instructions to monitor the association of pain and other symptoms with menstrual cycle changes, and planning for times in participants' menstrual cycles when symptoms might increase. Participant contacts were timed according to each participant's menstrual cycle.
- Continuous Oral Contraceptives: 20 mcg ethinyl estradiol and 100 mcg levonorgestrel Combination pill (20 mcg ethinyl estradiol and 100 mcg levonorgestrel) taken daily for 6 months.
Period: Treatment
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives
Started | 60 | 57 | 74
Completed | 54 | 50 | 36
Not Completed | 6 | 7 | 38
Not completed — Became ineligible post-randomization | 0 | 1 | 16
Not completed — Moved out of state | 1 | 1 | 1
Not completed — Completed no treatment | 5 | 5 | 21
Period: Short Term (6 Month) Follow up
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives
Started | 59 (Greater than number completing treatment: intent to treat analysis) | 55 (Greater than number completing treatment: intent to treat analysis) | 57 (Greater than number completing treatment: intent to treat analysis)
Completed | 50 | 47 | 46
Not Completed | 9 | 8 | 11
Not completed — Lost to Follow-up | 9 | 8 | 11
Period: Long Term (12 Month) Follow up
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives
Started | 59 (Greater than number completing treatment: intent to treat analysis) | 55 (Greater than number completing treatment: intent to treat analysis) | 57 (Greater than number completing treatment: intent to treat analysis)
Completed | 48 | 46 | 48
Not Completed | 11 | 9 | 9
Not completed — Lost to Follow-up | 11 | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives | Total
Number analyzed (Participants) | 51 | 47 | 49 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 47 | 49 | 147
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.1 (7.4) | 25.4 (5.7) | 28.6 (6.9) | 27.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 47 | 49 | 147
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 47 | 49 | 147

OUTCOME MEASURES:

1. Primary Outcome: Characteristic Pain Intensity (Characteristic Intensity of Facial Pain)
Description: Average of 0-10 ratings of current facial pain, average facial pain in the last month and worst facial pain in the last month, where 0 is no pain and 10 is pain as bad as could be. For the combined outcome, the minimum score is 0 and maximum is 10, with 0 being better (no pain) and 10 being the worst outcome.
Time Frame: 6 months
Population: Participants with 6 month follow up data. Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives
Number analyzed (Participants) | 50 | 47 | 46
units on a scale | 3.1 (1.8) | 2.9 (2.0) | 3.6 (2.2)
Statistical Analysis 1: Comparison: Self Management vs Targeted Self Management vs Continuous Oral Contraceptives; The null hypothesis was that mean characteristic pain intensity at 6-month follow up is equal across the three groups; Test type: Superiority or Other; p = 0.19, Regression, Linear; Linear regression was used to compare group means at follow up, adjusted for baseline values of the outcome variable

2. Secondary Outcome: Number of Participants With Pain-Related Activity Interference
Description: Degree to which pain interferes with: daily activities, work and household activities, recreational activities (mean of 3 0-10 ratings); dichotomized as presence/absence of pain-related activity interference
Time Frame: 6 Months
Population: Participants with 6 month follow up data. Intention to treat analysis.
Measure: Number; unit: participants
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives
Number analyzed (Participants) | 50 | 47 | 46
participants | 21 | 19 | 25
Statistical Analysis 1: Comparison: Self Management vs Targeted Self Management vs Continuous Oral Contraceptives; Test type: Superiority or Other; p = 0.27, Regression, Logistic; Adjusted for baseline value of the outcome variable

3. Primary Outcome: Characteristic Pain Intensity (Characteristic Intensity of Facial Pain)
Description: as for outcome 1
Time Frame: 12 months
Population: Participants with 12 month follow up data. Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives
Number analyzed (Participants) | 48 | 46 | 48
Units on a scale | 2.8 (1.6) | 2.8 (2.0) | 3.9 (1.9)
Statistical Analysis 1: Comparison: Self Management vs Targeted Self Management vs Continuous Oral Contraceptives; The null hypothesis was that mean characteristic pain intensity at 12-month follow up is equal across the three groups; Test type: Superiority or Other; p = 0.003, Regression, Linear; Group means compared with linear regression adjusted for baseline values. Adjusted difference: -1.0 between SMT and COCT, -1.0 between TSMT and COCT

4. Secondary Outcome: Number of Participants With Pain-Related Activity Interference
Description: as for outcome 2
Time Frame: 12 months
Population: Participants with 12 month follow up data. Intention to treat analysis.
Measure: Number; unit: participants
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives
Number analyzed (Participants) | 48 | 46 | 48
participants | 19 | 17 | 30
Statistical Analysis 1: Comparison: Self Management vs Targeted Self Management vs Continuous Oral Contraceptives; Test type: Superiority or Other; p = 0.016, Regression, Logistic; Adjusted for baseline value of the outcome variable

ADVERSE EVENTS:
Time Frame: Treatment period (6 months, all groups) and 2 months after treatment for continuous oral contraceptive group.
Description: Subjects in the continuous oral contraceptive group were told to report any problems to the nurse practitioner.
Arm/Group | Self Management | Targeted Self Management | Continuous Oral Contraceptives
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/50 | 0/36
Other Adverse Events (participants affected / at risk) | 0/54 | 0/50 | 23/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self Management (N=54) | Targeted Self Management (N=50) | Continuous Oral Contraceptives (N=36)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) — Expected adverse event with use of oral contraceptives
Breakthrough bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 17 (20) — Expected event with onset of use of continuous oral contraceptives
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) — Expected event with use of oral contraceptives
Cramping (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) — Expected event with use of oral contraceptives
Headaches (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) — Expected event with use of oral contraceptives
Moodiness/increased emotionality (General disorders) | 0 (0) | 0 (0) | 3 (3)
Weight gain (General disorders) | 0 (0) | 0 (0) | 2 (2) — Expected event with use of oral contraceptives

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No